CLINICAL TRIAL: NCT03488420
Title: Canadian EdoxAban (Lixiana®) Registry in Patients With ATrial Fibrillation and/or ATrial Flutter With Confirmed ValvUlar HeaRt DiseasE (CAPTURE)
Brief Title: Canadian EdoxAban(Lixiana®) Registry in Patients With ATrial Fibrillation/Flutter With Confirmed ValvUlar HeaRt DiseasE
Acronym: CAPTURE
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Other Study IDs: MHICC-2017-001
Record Dates: First submitted 2018-03-20; First posted 2018-04-05 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation and Flutter; Valvular Heart Disease
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial Fibrillation and/or Atrial Flutter: Subjects taking edoxaban 30mg or 60 mg will be followed for 2 years. Subjects will perform the Montreal Cognitive Assessment (MoCA) Test at baseline and 1-year follow up. They will also answer the Anti-Clot Treatment questionnaire (ACTS-Q) at 1-year.
  Interventions: Drug: Edoxaban Pill

INTERVENTIONS:
Drug: Edoxaban Pill — Subjects will be taking edoxaban 30 or 60 mg
  Other Names: Lixiana; edoxaban tosylate monhydrate

SUMMARY:
The objective of this registry is the characterization of patients with atrial fibrillation (AF) and/ or atrial flutter (AFL) with confirmed VHD who are prescribed edoxaban in a real life clinical setting.

DETAILED DESCRIPTION:
This is an observational, prospective, multicenter, edoxaban Canadian registry of adults (≥18) diagnosed or confirmed with AF and/or AFL with VHD, within the last 12 months, according to local standard procedures and judged by the investigator to be at risk of stroke and in whom anticoagulation with NOAC is clinically indicated and who are prescribed edoxaban. A total of about 300 patients will be enrolled from approximately 10 sites in Quebec. Patients will be treated according to standard local practices. There is no formal interventions. Treatment decisions are left to the physician's discretion.

Registry data will be collected by the investigator or delegate at baseline, 6, 12 and 24 months and recorded in the electronic Case Report Form (eCRF).

Data available in the patient's file will be collected. The only procedure to be performed in the context of this registry is the completion of questionnaires: the Montreal Cognitive Assessment (MoCA©) test and the Anti-Clot-Treatment Scale (ACTS-Q) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 18 years at baseline (signing of consent);
2. Willing and able to provide written informed consent;
3. Patient diagnosed or confirmed with AF and/or AFL within the last 12 months of signed consent form;
4. Patient with VHD confirmed by echocardiography within the last 36 months of signed consent form except for mitral stenosis that must be confirmed within the last 12 months;
5. Patient at risk for stroke in whom a long term oral anticoagulation is indicated and who are prescribed edoxaban.

Exclusion Criteria:

1. Patients with AF and/or AFL secondary to reversible cause;
2. Patients with a mechanical heart valve or rheumatic mitral stenosis, or moderate and severe non rheumatic mitral stenosis;
3. Patients planned to have an intervention for valvular heart disease in the next 12 months;
4. Pregnant or breastfeeding women.
5. Short term anticoagulation post cardioversion or ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed or confirmed with Atrial Fibrillation (AF) and/or atrial flutter (AFL) with valvular heart disease (VHD) within the last 12 months, according to local standard procedures, judged by the investigator to be at risk of stroke and in whom anticoagulation with a NOAC drugs is clinically indicated and who are prescribed edoxaban.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Characterization of patients with diagnosed or confirmed atrial fibrillation (AF) and/or atrial flutter (AFL) with valvular heart disease (VHD), within the last 12 months | 2 years
Patient treatment satisfaction using Anti-Clot Treatment Scale (ACTS) | 2 years
Cognitive function using the Montreal Cognitive Assessment (MoCA) test | 2 years
Compliance of subjects to edoxaban treatment | 2 years
Reasons for choosing edoxaban and reasons for the dosage | 2 years
Percentage of patients on appropriate dosage of edoxaban (60 mg and 30 mg if dose reduction criteria) | 2 years
Stroke (hemorrhagic stroke, ischemic stroke), transient ischemic attack (TIA) and systemic embolism events (SEE) | 2 years
Bleeding (Frequency, Location, Severity, Type of intervention and Outcome) | 2 years
Death (CV and non-CV) | 2 years
Adverse events (AEs) and serious adverse events (SAEs) related to edoxaban | 2 years
Physician satisfaction with regards to edoxaban treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katia Dyrda, MD, Principal Investigator — Montreal Heart Institute
Locations (9):
- Canada (9):
  - CIUSSS de l'Estrie-CHUS-Centre Haute-Yamaska-hôpital de Granby, Granby, Quebec
  - CISSS de la Montérégie Centre, Greenfield Park, Quebec
  - CISSS de Laval, Laval, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - IUCPQ, Québec, Quebec
  - CISSS du Bas-Saint-Laurent/Hôpital Régional de Rimouski, Rimouski, Quebec
  - CISSS de Chaudière-Appalaches - Hopital Saint-Georges, Saint-Georges, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - CIUSSS de la Mauricie-et-du-Centre-du-Québec, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No